CLINICAL TRIAL: NCT04219059
Title: MR Radiomic Features in Prostate Cancer
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: IBFM-CNR (Istituto di Bioimmagini e Fisiologia Molecolare, National Research Council, Segrate, Italy (Unknown)
Responsible Party: Principal Investigator, Francesco De Cobelli, Head, Radiology Department, IRCCS San Raffaele
Other Study IDs: ProTex
Record Dates: First submitted 2019-12-25; First posted 2020-01-06 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Prostate Cancer
Keywords: cancer; prostate; radiomics; MRI; prognostic factors
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A combination of correct interpretation of imaging and biopsy has given promising results in terms of detecting clinically significant cancer at radical prostatectomy.

DETAILED DESCRIPTION:
Quantitative approaches to medical image analysis have been developed in recent years with the aim to overcome the limitation of qualitative image interpretation, and provide biomarkers for disease characterization. In particular, the new paradigm, "radiomics", is emerging as the high-throughput extraction of quantitative features from imaging which can aid in characterizing phenotype as in vivo expression of tumoral genotype. The goal of radiomics is to extract accurate and reliable quantitative biomarkers which enhance diagnostic confidence in oncology. A combination of correct interpretation of imaging and biopsy has given promising results in terms of detecting clinically significant cancer at radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* In house MRI with contrast medium
* PCa (prostate cancer) biopsy proven diagnosis
* In house radical prostatectomy

Exclusion Criteria:

* < 18 years of age
* MRI without contrast medium
* Radical prostatectomy executed not in Institution

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: 200 male patients who have a pre-intervention prostate MRI with contrast agent from December 2015 to August 30, 2019 and biopsy proven Pca diagnosis, followed by radical prostatectomy will be evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Number of surrogate bioimaging markers of histological characteristics in MR images | 0-2 years
  Segment tumor volumes on the ADC map and extract different imaging features

SECONDARY OUTCOMES:
Radiomic features from MRI | 0-2 years
  Evaluate if radiomic features on primitive prostate lesions can describe lymph node involvement.
Extract radiomic features | 0-2 years
  Evaluate if radiomic features fro MRIon primitive prostate lesions can describe disease extension.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy